CLINICAL TRIAL: NCT04277754
Title: Correspondence Between Motor and Road Development in 2-year-old Children With Typical Development
Brief Title: Motor and Visual Development in 2 Year Olds
Status: Completed | Type: Observational
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Elena Piñero Pinto, Principal investigator, University of Seville
Other Study IDs: Development
Record Dates: First submitted 2020-01-09; First posted 2020-02-20 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Development, Child; Motor Skills Disorders; Visual Disorder
Keywords: developmet; motor; visual; infant
MeSH Terms: conditions — Motor Skills Disorders; Vision Disorders | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- two-year-old children with typical development
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — To Observe and describe motor and visual development

SUMMARY:
It is a study where investigators are going to measure variables related to motor development and vision through objective tests in children with typical development of two years of age.

ELIGIBILITY:
Inclusion Criteria:

* typical development
* be enrolled in a nursery school of the University of Seville

Exclusion Criteria:

* visual deficit
* developmental disorder

Ages: 24 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: two-year-old children with typical development
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Motor development | Up to two weeks
  Researchers will use objective tests to measure the equivalent age of development in this area with respect to their chronological age and the percentage of skills acquired in the different dimensions of the motor area.
  The evidence that will be used will be for this purpose will be:
  - Peabody Developmental Motor Scales- II.
  It will take about 15 minutes of evaluation where the child will be asked to reproduce a series of general body movements, as well as some hand and object skills
Motor development | Up to two weeks
  Researchers will use objective tests to measure the coefficients of development in this area with respect to their chronological age and the percentage of skills acquired in the different dimensions of the motor area.
  The evidence that will be used will be for this purpose will be:
  - Peabody Developmental Motor Scales- II.
  It will take about 15 minutes of evaluation where the child will be asked to reproduce a series of general body movements, as well as some hand and object skills

SECONDARY OUTCOMES:
Visual acuity | Up to two weeks
  Researchers will check visual acuity through the Cardif Test. It is non-invasive and the collaboration required by the child is minimal.
Visual axis alignment | Up to two weeks
  Researchers will check visual axis alignment throught the Cover Test. It Is non-invasive and the collaboration required by the child is minimal.
Three dimensional vision capability | Up to two weeks
  Researchers will check three-dimensional vision capability throught the Lang Test. It is non-invasive and the collaboration required by the child is minimal.

CONTACTS AND LOCATIONS:
Locations (1):
- Elena Piñero Pinto, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided